CLINICAL TRIAL: NCT04213092
Title: "Single Setting ERCP and Laparoscopic Cholecystectomy is a Safe Procedure in Patients With Cholecysto-Choledocholithiasis: A Prospective Study in a Peripheral-Level Hospital"
Brief Title: Single Setting ERCP and Laparoscopic Cholecystectomy is a Safe Procedure in Patients With Cholecysto-Choledocholithiasis
Status: Completed | Type: Observational
Sponsor: Lumbini Medical College (Other)
Responsible Party: Principal Investigator, NabinPokharel, Ass. Prof. Dr Nabin Pokharel, Lumbini Medical College
Other Study IDs: IRC-LMC 01-H-015
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Choledocholithiasis With Cholecystitis With Obstruction; Choledocholithiasis With Acute and Chronic Cholecystitis; Cholelithiasis With Acute and Chronic Cholecystitis
Keywords: Common bile duct stones; Endoscopic Retrograde Cholangiopancreatography; Laparoscopic Cholecystectomy; Open Cholecystectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERCP+LC: Patients in this group underwent 2-stage ERCP+LC in a single setting. And, it was compared with our control group
  Interventions: Procedure: ERCP+LC
- OC+CBD: This group with 2-stage OC+CBD exploration in a single setting approach was taken as a control group.
  Interventions: Procedure: OC+CBD

INTERVENTIONS:
Procedure: ERCP+LC — Patients in this group underwent a single setting ERCP and Laparoscopic cholecystectomy.
  Groups: ERCP+LC
Procedure: OC+CBD — Patients in this group underwent a single setting open cholecystectomy and open CBD exploration.
  Groups: OC+CBD

SUMMARY:
The ideal management of cholecysto-choledocholithiasis is an open cholecystectomy (OC) with the common bile duct (CBD) exploration worldwide. The single setting 2-stage approach- endoscopic retrograde cholangiopancreatography (ERCP), endoscopic sphincterotomy (EST), and CBD clearance followed by laparoscopic cholecystectomy (LC) offers an advantage, mainly by reducing the hospital stay, the cost, and the morbidity. Investigators did a prospective study in patients admitted for the management of the cholecysto-choledocholithiasis in the Department of Surgery at the Lumbini Medical College and Teaching Hospital from November 2012- October 2015. They underwent 2-stage ERCP+LC in a single setting and investigators compared them with 2-stage OC+CBD exploration in a single setting approach. The patients with the open procedure were the investigator's control groups. All the included cases in the study were elective.

DETAILED DESCRIPTION:
This was a prospective study done on patients admitted for management of the cholecysto-choledocholithiasis in the Department of Surgery at the Lumbini Medical College and Teaching Hospital from November 2012 - October 2015. This is a peripheral setting hospital located in a remote city of Nepal-"Palpa". The study was approved by the institutional ethical committee- "IRC of Lumbini Medical College and Teaching Hospital" and written consent was obtained from all of the patients. A comprehensive literature search published in English was done till 2019 using Hinari, PubMed, Cochrane Library, EMBASE, Web of Science, and ScienceDirect.

This is an interim analysis of 160 patients with 83 (51.9%) patients in ERCP+LC and 77 (48.1%) in open procedure (OC with CBD exploration) group respectively. The primary objective was to compare the single setting ERCP+LC with OC+CBD exploration and the secondary objectives were to study 1) the feasibility of the procedure, 2) detect the morbidity (cholangitis, pancreatitis, abdominal collection, and wound infection), 3) the length of stay, and ). The stone clearance respectively. The investigators defined their single-setting procedure as ERCP followed by LC. The patients from an open procedure group were those who underwent the procedure before our team was trained to carry out the ERCP. This open procedure group also included 10 patients who underwent open surgery due to unsuccessful ERCP. And finally, investigators compared ERCP+LC group with those who underwent the open procedure. The inclusion and exclusion criteria for ERCP+LC and open procedure are shown in Table 1 and Table 2 respectively.

After being informed about the related therapeutic maneuver, the patients were chosen for the sequence of endoscopic procedures and LC. And, the unsuccessful patients underwent through the OC with CBD exploration along with choledochoscopy. General anesthesia with nasal endotracheal intubation was done in all the patients. Antibiotic prophylaxis was given according to the standard recommendation for cholecystectomy.18 The ERCP procedure was performed with the patients in the prone position. A duodenoscope (TJF160R, Fujinon, Japan) was inserted into the second segment of duodenum via the mouth. A cholangiogram was carried out using C-arm X-ray (SIEMENS) and an EST was performed to extract the CBD stones. The stones were removed by basket or balloon catheter. Stones larger than 10 mm were removed using a mechanical lithotripter. Following ERCP, care was taken to remove all the gas from the stomach to facilitate LC. The patients were then placed in the reverse Trendelenburg position. LC was performed using the four trocar technique. A sub-hepatic drain was positioned if there was any concern about the possible bile leakage or bleeding in the postoperative period.

In cases of failed ERCP, the patients were placed in the supine position and OC with CBD explorations were performed in the same setting. A right subcostal incision was given for the open surgery. Cholecystectomy was performed ante-grade or retro-grade technique depending upon the anatomical variations of the gallbladder. CBD was opened below the opening of the cystic duct and stone clearances were done. To assure the stone clearances intraoperative choledochoscopies were performed. All the procedure viz. ERCP, LC, and open surgeries were performed by an experienced single surgeon and his team.

The statistical data were analyzed with a t-test, Pearson's χ2, Fisher's exact test, Mann Whitney's test, and Kruskal Wallis test using a statistical analysis program (SPSS 16), p <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. All the sonological proven cases of choledocholithiasis with cholelithiasis.
2. CBD diameter <2cm.
3. Age >13 yrs.

Exclusion Criteria:

1. Clinical, radiologic, or biochemical evidence of cholangitis and pancreatitis.
2. Evidence of cirrhosis, intrahepatic gallbladder, liver mass or abscess, neoplasm, Suppurative or necrotizing cholecystitis, gall bladder empyema, or perforation, Pregnancy.

Age >85 yrs.

Ages: 13 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was carried out in a peripheral setting hospital located in a remote city of Nepal-"Palpa" and the population is heterogeneous in terms of age.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Compare ERCP+LC with OC+CBD exploration | 7 days
  To compare the single setting ERCP+LC with OC+CBD exploration and the Feasibility of the procedure at the peripheral setting hospital.

SECONDARY OUTCOMES:
Morbidity | 7 days
  Detect cholangitis, pancreatitis, abdominal collection, and wound infection respectively
Length | 7 days
  The length of Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Chet R Pant, MD, MPH, Study Chair — Lumbini Medical College & Teaching Hospital Ltd, Kathmandu University

IPD SHARING:
Plan to Share IPD: Yes
We can share our study IPD to interested researchers. Please email us at nabin.pokharel@gmail.com
Time Frame: Data will be available for all interested researchers via the publication.
Access Criteria: interested researchers in the field of ERCP; Laparoscopic Cholecystectomy; Open Cholecystectomy, Laparoscopic CBD Exploration, Open CBD Exploration.

REFERENCES:
- [Background] European Association for the Study of the Liver (EASL). Electronic address: easloffice@easloffice.eu. EASL Clinical Practice Guidelines on the prevention, diagnosis and treatment of gallstones. J Hepatol. 2016 Jul;65(1):146-181. doi: 10.1016/j.jhep.2016.03.005. Epub 2016 Apr 13. No abstract available. PMID 27085810
- [Background] Zhu HY, Xu M, Shen HJ, Yang C, Li F, Li KW, Shi WJ, Ji F. A meta-analysis of single-stage versus two-stage management for concomitant gallstones and common bile duct stones. Clin Res Hepatol Gastroenterol. 2015 Oct;39(5):584-93. doi: 10.1016/j.clinre.2015.02.002. Epub 2015 Apr 27. PMID 25936687
- [Background] ASGE Standards of Practice Committee; Maple JT, Ikenberry SO, Anderson MA, Appalaneni V, Decker GA, Early D, Evans JA, Fanelli RD, Fisher D, Fisher L, Fukami N, Hwang JH, Jain R, Jue T, Khan K, Krinsky ML, Malpas P, Ben-Menachem T, Sharaf RN, Dominitz JA. The role of endoscopy in the management of choledocholithiasis. Gastrointest Endosc. 2011 Oct;74(4):731-44. doi: 10.1016/j.gie.2011.04.012. No abstract available. PMID 21951472
- [Background] Gurusamy KS, Giljaca V, Takwoingi Y, Higgie D, Poropat G, Stimac D, Davidson BR. Ultrasound versus liver function tests for diagnosis of common bile duct stones. Cochrane Database Syst Rev. 2015 Feb 26;2015(2):CD011548. doi: 10.1002/14651858.CD011548. PMID 25719223
- [Background] Miletic D, Uravic M, Mazur-Brbac M, Stimac D, Petranovic D, Sestan B. Role of magnetic resonance cholangiography in the diagnosis of bile duct lithiasis. World J Surg. 2006 Sep;30(9):1705-12. doi: 10.1007/s00268-005-0459-1. PMID 16850153
- [Background] Freitas ML, Bell RL, Duffy AJ. Choledocholithiasis: evolving standards for diagnosis and management. World J Gastroenterol. 2006 May 28;12(20):3162-7. doi: 10.3748/wjg.v12.i20.3162. PMID 16718834
- [Background] Lee A, Min SK, Park JJ, Lee HK. Laparoscopic common bile duct exploration for elderly patients: as a first treatment strategy for common bile duct stones. J Korean Surg Soc. 2011 Aug;81(2):128-33. doi: 10.4174/jkss.2011.81.2.128. Epub 2011 Aug 3. PMID 22066112
- [Background] Gurusamy KS, Giljaca V, Takwoingi Y, Higgie D, Poropat G, Stimac D, Davidson BR. Endoscopic retrograde cholangiopancreatography versus intraoperative cholangiography for diagnosis of common bile duct stones. Cochrane Database Syst Rev. 2015 Feb 26;2015(2):CD010339. doi: 10.1002/14651858.CD010339.pub2. PMID 25719222
- [Background] Gomez-Torres GA, Gonzalez-Hernandez J, Lopez-Lizarraga CR, Navarro-Muniz E, Ortega-Garcia OS, Bonnet-Lemus FM, Abarca-Rendon FM, De la Cerda-Trujillo LF. Intraoperative cholangiography versus magnetic resonance cholangiography in patients with mild acute biliary pancreatitis: A prospective study in a second-level hospital. Medicine (Baltimore). 2018 Nov;97(44):e12976. doi: 10.1097/MD.0000000000012976. PMID 30383648
- [Background] Alexakis N, Connor S. Meta-analysis of one- vs. two-stage laparoscopic/endoscopic management of common bile duct stones. HPB (Oxford). 2012 Apr;14(4):254-9. doi: 10.1111/j.1477-2574.2012.00439.x. Epub 2012 Feb 3. PMID 22404264
- [Background] ElGeidie AA, ElShobary MM, Naeem YM. Laparoscopic exploration versus intraoperative endoscopic sphincterotomy for common bile duct stones: a prospective randomized trial. Dig Surg. 2011;28(5-6):424-31. doi: 10.1159/000331470. Epub 2012 Jan 7. PMID 22236538